CLINICAL TRIAL: NCT02706457
Title: Do Improvements in Functionality on the ICU Give a Reduction of Post Intensive Care Syndrome
Brief Title: Post Intensive Care Syndrome
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Other Study IDs: nWMO 143
Record Dates: First submitted 2016-02-16; First posted 2016-03-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Post Intensive Care Syndrome; Barthel Index
Keywords: intensive care; functionality
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort 2012 - 2014: all patients admitted for > 48 hours on the Intensive Care Unit in 2012, 2013 and 2014
  Interventions: Other: Barthel index for functionality

INTERVENTIONS:
Other: Barthel index for functionality — The Barthel Index for functionality is done standard in all patients after intensive care admission

SUMMARY:
Barthel Index and demographic variables of patients were collected to investigate the question whether the improvements of the functionality improves the Barthel Index over the years.

DETAILED DESCRIPTION:
idem

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* length of stay longer than 48 hours

Exclusion Criteria:

* no exclusion criteria if inclusion is correct

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated in Intensive Care for minimal 48 hours, during the years 2012 - 2014
Sampling Method: Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Difference in Barthel Index | from januari 2012 until decembre 2014
  barthel index is analyzed over the years 2012 - 2014

SECONDARY OUTCOMES:
Relation between Barthel Index and length of stay in ICU | from januari 2012 until decembre 2014

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — MCL
Locations (1):
- Medical Center Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No